CLINICAL TRIAL: NCT02029443
Title: A Phase 1/2, Multicenter, Open-label, and Dose-escalation Study of ACP-196 in Subjects With Chronic Lymphocytic Leukemia, Richter's Syndrome or Prolymphocytic Leukemia
Brief Title: ACP-196 (Acalabrutinib), a Novel Bruton Tyrosine Kinase (BTK) Inhibitor, for Treatment of Chronic Lymphocytic Leukemia, Richter's Syndrome or Prolymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACE-CL-001; 2023-509346-35-00 (Registry Identifier: CTIS(EU)); 2014-000440-15 (EudraCT Number)
Record Dates: First submitted 2014-01-06; First posted 2014-01-08 (Estimated); Results first posted 2022-09-10 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Richter's Syndrome; Prolymphocytic Leukemia
Keywords: Bruton's tyrosine kinase inhibitor
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Prolymphocytic | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Relapsed/Refractory Cohort (Experimental): Phase 1 (dose-escalation) and Phase 2 (dose-expansion) will be conducted for participants with relapsed/refractory CLL or SLL. In Phase 1, participants will receive oral once daily (QD) acalabrutinib at Dose 1 (Cohort 1), Dose 2 (Cohort 2a), Dose 3 (Cohort 3), and Dose 4 (Cohort 4a), and twice daily (BID) acalabrutinib at Dose 1 (Cohort 2b) and Dose 5 (Cohort 4b) for 28 days (1 cycle). In Phase 2, participants will receive oral acalabrutinib at Dose 1 BID (Cohort 2b) or Dose 5 QD (Cohort 2c, later will be switched to Dose 1 BID per protocol amendment 6) until disease progression or until the investigator will consider the study treatment to be intolerable or no longer in the participant's best interest. Participants from Phase 1 will be continued to receive Dose 1 BID until disease progression or until the investigator will consider the study treatment to be intolerable or no longer in the participant's best interest.
  Interventions: Drug: Acalabrutinib
- Treatment-naive Cohort (Experimental): Treatment-naïve participants with confirmed CLL or SLL, will receive oral acalabrutinib Dose 5 QD (Cohort 7, later will be switched to Dose 1 BID per protocol amendment 6) or Dose 1 BID (Cohort 11) until disease progression or until the investigator will consider the study treatment to be intolerable or no longer in the participant's best interest.
  Interventions: Drug: Acalabrutinib
- Ibrutinib-intolerant Cohort (Experimental): Participants with confirmed CLL or SLL and were not tolerating ibrutinib treatment, will receive oral acalabrutinib Dose 5 QD (Cohort 8a, later switched to Dose 1 BID per protocol amendment 4) or Dose 1 BID (Cohort 8b) until disease progression or until the investigator will consider the study treatment to be intolerable or no longer in the participant's best interest.
  Interventions: Drug: Acalabrutinib
- Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort (Experimental): Participants with diffuse large B-cell lymphoma (DLBCL) Richter's transformation (RS) or prolymphocytic leukemia (PLL) transformation, will receive oral acalabrutinib Dose 5 BID (Cohort 9) until disease progression or until the investigator will consider the study treatment to be intolerable or no longer in the participant's best interest.
  Interventions: Drug: Acalabrutinib
- Ibrutinib Relapsed/Refractory Cohort (Experimental): Participants with confirmed CLL/SLL and had relapsed/refractory to ibrutinib treatment, will receive oral acalabrutinib Dose 5 QD (Cohort 10) until disease progression or until the investigator will consider the study treatment to be intolerable or no longer in the participant's best interest.
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — Participants will receive acalabrutinib as stated in the arms' description.
  Other Names: ACP-196

SUMMARY:
This study is evaluating the safety and efficacy of a new BTK inhibitor, acalabrutinib, for the treatment of chronic lymphocytic leukemia (CLL)/small lymphocytic lymphoma (SLL).

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age with a confirmed diagnosis of CLL/SLL, which has relapsed after, or been refractory to, ≥ 2 previous treatments for CLL/SLL.
2. Must have measurable CLL/SLL defined as ≥ 1 lymph node ≥ 2 cm as measured in the longest diameter.
3. Active disease meeting ≥ 1 of the following International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 criteria for requiring treatment:

   1. Evidence of progressive marrow failure as manifested by the development of, or worsening of, anemia (hemoglobin < 10 g/dL) and/or thrombocytopenia (platelets < 100,000/μL).
   2. Massive (i.e., ≥ 6 cm below the left costal margin), progressive, or symptomatic splenomegaly.
   3. Massive nodes (i.e., ≥ 10 cm in the longest diameter), progressive, or symptomatic lymphadenopathy.
   4. Progressive lymphocytosis with an increase of > 50% over a 2-month period or a lymphocyte doubling time (LDT) of < 6 months. The LDT may be obtained by linear regression extrapolation of absolute lymphocyte counts (ALC) obtained at intervals of 2 weeks over an observation period of 2 to 3 months. In participants with initial blood lymphocyte counts of < 30 X 10^9/L (30,000/μL), LDT should not be used as a single parameter to define indication for treatment. In addition, factors contributing to lymphocytosis or lymphadenopathy other than CLL (eg, infections) should be excluded.
   5. Autoimmune anemia and/or thrombocytopenia that is poorly responsive to standard therapy.
   6. Constitutional symptoms documented in the participant's chart with supportive objective measures, as appropriate, defined as ≥ 1 of the following disease-related symptoms or signs:

   i. Unintentional weight loss ≥ 10% within the previous 6 months before screening.

   ii. Fevers higher than 100.5°F or 38.0°C for 2 or more weeks before screening without evidence of infection.

   iii. Night sweats for > 1 month before screening without evidence of infection.
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
5. Agreement to use highly effective methods of contraception during the study and for 2 days after the last dose of study drug if sexually active and able to bear or beget children (see Section 3.7.9 for list of highly effective methods of contraception).
6. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
7. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (in accordance with national and local participant privacy regulations).

Inclusion Criteria for Treatment Subgroups

1. Treatment Naive only: Men and women ≥ 18 years of age with confirmed diagnosis of CLL/SLL, who require treatment per National Cancer Institute (NCI) or International Working Group guidelines and a) do not want to receive chemoimmunotherapy or b) have comorbidities that would preclude chemoimmunotherapy.
2. Ibrutinib Intolerant only: Men and women ≥ 18 years of age with confirmed diagnosis of CLL/SLL who are not tolerating ibrutinib due to ibrutinib-related AEs.
3. Richter's Syndrome/Prolymphocytic Leukemia Transformation only: Men and women ≥ 18 years of age and biopsy proven diffuse large B cell lymphoma (DLBCL) Richter's transformation or prolymphocytic leukemia transformation.
4. Ibrutinib relapsed/refractory (R/R) only: Men and women ≥ 18 years of age with confirmed diagnosis of CLL/SLL whose best response after 2 cycles of ibrutinib therapy was stable disease or nonresponse or who initially responded to ibrutinib therapy and now have signs of clinical progression.

Exclusion Criteria:

1. Prior malignancy, except for adequately treated basal cell, squamous cell skin cancer or in situ cervical cancer. Participants with other prior malignancies from which the participant has been disease free for ≥ 2 years may be included if approved by the medical monitor.
2. A life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the participant's safety, interfere with the absorption or metabolism of acalabrutinib, or put the study outcomes at undue risk.
3. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or left ventricular ejection fraction (LVEF) ≤ 40%.
4. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
5. Any immunotherapy within 4 weeks of first dose of study drug.
6. For participants with recent chemotherapy or experimental therapy the first dose of study drug must occur after 5 times the half-life of the agent(s).
7. Relapsed after, or refractory to, prior BTK inhibitor therapy (Note: Does not apply to Ibrutinib R/R or Richter's Syndrome Group).
8. Any history of Richter's transformation (Note: Does not apply to Richter's Syndrome Group).

10. Central nervous system (CNS) involvement by lymphoma. 11. Grade ≥ 2 toxicity (other than alopecia) continuing from prior anticancer therapy including radiation.

12. Known history of human immunodeficiency virus (HIV) or serologic status indicating active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection or any uncontrolled active systemic infection. Participants with hepatitis B core antibody positive who are surface antigen negative or who are hepatitis C antibody positive will need to have a negative polymerase chain reaction (PCR) result before enrollment. Those who are hepatitis B surface antigen positive or hepatitis B PCR positive and those who are hepatitis C PCR positive will be excluded.

13. Uncontrolled autoimmune hemolytic anemia (AIHA) or immune thrombocytopenic purpura (ITP) defined as declining hemoglobin or platelet count secondary to autoimmune destruction within the screening period or requirement for high doses of steroids (> 20 mg daily of prednisone daily or equivalent).

14. History of stroke or intracranial hemorrhage within 6 months prior to the first dose of study drug.

15. Requires treatment with proton-pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole).

16. Requires anticoagulation with warfarin or equivalent vitamin K antagonists (eg, phenprocoumon) within 7 days of first dose of study drug.

17. Major surgery within 4 weeks before first dose of study drug. 18. ANC < 0.75 x 10^9/L or platelet count < 50 x 10^9/L unless there is bone marrow involvement.

19. Total bilirubin > 1.5 x upper limit of normal (ULN) (total bilirubin ≤ 2.5 x ULN allowed in participants with autoimmune hemolytic anemia that is otherwise controlled); and aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3.0 x ULN unless disease related.

20. Serum amylase > 1.5 x ULN or serum lipase > 1.5 x ULN. 21. Significant screening electrocardiogram (ECG) abnormalities including, 2nd degree AV block type II, 3rd degree block, Grade 2 or higher bradycardia, or QTc ≥ 480 ms.

22. Cardiac troponin I levels above the limit of normal as specified by the manufacturer.

23. Breast feeding or pregnant. 24. History of bleeding diathesis (eg, hemophilia, von Willebrand disease). 25. Concurrent participation in another therapeutic clinical trial. 26. Estimated creatinine clearance of < 30 mL/min, calculated using the formula of Cockcroft and Gault [(140-Age) • Mass (kg)/(72 • creatinine mg/dL); multiply by 0.85 if female].

27. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2014-01-30 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2027-06-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613 acertamc@dlss.com
Locations (12):
- United States (8):
  - Research Site, Boston, Massachusetts
  - Research Site, New Hyde Park, New York
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Fort Worth, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
- Research Site, Milan, Italy
- United Kingdom (3):
  - Research Site, Leeds
  - Research Site, London
  - Research Site, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Nuttall B, Karl DL, Burke K, Callahan M, Mendler K, Cingolani P, Criscione S, Naumenko S, Bibikova E, Munugalavadla V, Byrd JC, Furman RR, Brown JR, Mortlock A, Dougherty BA, Carl Barrett J, Scaltriti M, Hadfield J. Comprehensive comparison of enzymatic and bisulfite DNA methylation analysis in clinically relevant samples. Clin Epigenetics. 2025 Oct 3;17(1):156. doi: 10.1186/s13148-025-01959-0. PMID 41044668
- [Derived] Bibikova E, Parsa S, Floren M, Law B, Clevenger T, Cheung J, De Jesus G, Burke K, Gulrajani M, Yamaguchi K, Do P, Dougherty B, Whitston D, Brock G, Munugalavadla V, Frigault MM, Hartmann TN, Byrd JC, Furman RR, Brown JR, Covey T, Mortlock A. Molecular Profiling Identifies CD49d and CD79b as Predictive Markers for Acquired Acalabrutinib Resistance in Patients With Chronic Lymphocytic Leukemia. Hematol Oncol. 2025 Jan;43(1):e70008. doi: 10.1002/hon.70008. PMID 39716442
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886
- [Derived] Eyre TA, Schuh A, Wierda WG, Brown JR, Ghia P, Pagel JM, Furman RR, Cheung J, Hamdy A, Izumi R, Patel P, Wang MH, Xu Y, Byrd JC, Hillmen P. Acalabrutinib monotherapy for treatment of chronic lymphocytic leukaemia (ACE-CL-001): analysis of the Richter transformation cohort of an open-label, single-arm, phase 1-2 study. Lancet Haematol. 2021 Dec;8(12):e912-e921. doi: 10.1016/S2352-3026(21)00305-7. Epub 2021 Nov 1. PMID 34735860
- [Derived] Byrd JC, Wierda WG, Schuh A, Devereux S, Chaves JM, Brown JR, Hillmen P, Martin P, Awan FT, Stephens DM, Ghia P, Barrientos J, Pagel JM, Woyach JA, Burke K, Covey T, Gulrajani M, Hamdy A, Izumi R, Frigault MM, Patel P, Rothbaum W, Wang MH, O'Brien S, Furman RR. Acalabrutinib monotherapy in patients with relapsed/refractory chronic lymphocytic leukemia: updated phase 2 results. Blood. 2020 Apr 9;135(15):1204-1213. doi: 10.1182/blood.2018884940. PMID 31876911
- [Derived] Awan FT, Schuh A, Brown JR, Furman RR, Pagel JM, Hillmen P, Stephens DM, Woyach J, Bibikova E, Charuworn P, Frigault MM, Hamdy A, Izumi R, Linghu B, Patel P, Wang MH, Byrd JC. Acalabrutinib monotherapy in patients with chronic lymphocytic leukemia who are intolerant to ibrutinib. Blood Adv. 2019 May 14;3(9):1553-1562. doi: 10.1182/bloodadvances.2018030007. PMID 31088809
- [Derived] Long M, Beckwith K, Do P, Mundy BL, Gordon A, Lehman AM, Maddocks KJ, Cheney C, Jones JA, Flynn JM, Andritsos LA, Awan F, Fraietta JA, June CH, Maus MV, Woyach JA, Caligiuri MA, Johnson AJ, Muthusamy N, Byrd JC. Ibrutinib treatment improves T cell number and function in CLL patients. J Clin Invest. 2017 Aug 1;127(8):3052-3064. doi: 10.1172/JCI89756. Epub 2017 Jul 17. PMID 28714866
- [Derived] Byrd JC, Harrington B, O'Brien S, Jones JA, Schuh A, Devereux S, Chaves J, Wierda WG, Awan FT, Brown JR, Hillmen P, Stephens DM, Ghia P, Barrientos JC, Pagel JM, Woyach J, Johnson D, Huang J, Wang X, Kaptein A, Lannutti BJ, Covey T, Fardis M, McGreivy J, Hamdy A, Rothbaum W, Izumi R, Diacovo TG, Johnson AJ, Furman RR. Acalabrutinib (ACP-196) in Relapsed Chronic Lymphocytic Leukemia. N Engl J Med. 2016 Jan 28;374(4):323-32. doi: 10.1056/NEJMoa1509981. Epub 2015 Dec 7. PMID 26641137
- See also: Redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-001&attachmentIdentifier=8afe4e09-79d8-4dac-844d-3d25bed390c4&fileName=ACE-CL-001_SAP_redacted.pdf&versionIdentifier=
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-001&attachmentIdentifier=7e985bdb-edff-4078-b568-1f1eccac21c2&fileName=ACE-CL-001-CSP_redacted.pdf&versionIdentifier=
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-001&attachmentIdentifier=9bcc8806-9a38-4b54-9063-d7d514344c0f&fileName=ACE-CL-001-CSRsynopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 306 enrolled participates, 5 participants were not treated with the study drug. The data of "All treated population" was collected and analyzed. The results data are reported per the primary completion date (data cut-off date of 15Jul2021). There will be no updated results for all outcome measures at the time of end of study.
Groups:
- Relapsed/Refractory Cohort: Phase 1 (dose-escalation) and Phase 2 (dose-expansion) were conducted for participants with relapsed/refractory chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). In Phase 1, participants received oral once daily (QD) acalabrutinib at Dose 1 (Cohort 1), Dose 2 (Cohort 2a), Dose 3 (Cohort 3), and Dose 4 (Cohort 4a), and twice daily (BID) acalabrutinib at Dose 1 (Cohort 2b) and Dose 5 (Cohort 4b) for 28 days (1 cycle). In Phase 2, participants received oral acalabrutinib at Dose 1 BID (Cohort 2b) or Dose 5 QD (Cohort 2c, later switched to Dose 1 BID per protocol amendment 6) until disease progression or until the investigator considered the study treatment to be intolerable or no longer in the participant's best interest. Participants from Phase 1 continued to receive Dose 1 BID until disease progression or until the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Treatment-naive Cohort: Treatment-naïve participants with confirmed CLL or SLL, received oral acalabrutinib Dose 5 QD (Cohort 7, later switched to Dose 1 BID per protocol amendment 6) or Dose 1 BID (Cohort 11) until disease progression or until the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Ibrutinib-intolerant Cohort: Participants with confirmed CLL or SLL and were not tolerating ibrutinib treatment, received oral acalabrutinib Dose 5 QD (Cohort 8a, later switched to Dose 1 BID per protocol amendment 4) or Dose 1 BID (Cohort 8b) until disease progression or until the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort: Participants with diffuse large B-cell lymphoma (DLBCL) Richter's transformation (RS) or prolymphocytic leukemia transformation (PLL), received oral acalabrutinib Dose 5 BID (Cohort 9) until disease progression or until the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Ibrutinib Relapsed/Refractory Cohort: Participants with confirmed CLL/SLL and had relapsed/refractory to ibrutinib treatment, received oral acalabrutinib Dose 5 QD (Cohort 10) until disease progression or until the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
Period: Overall Study
Arm/Group | Relapsed/Refractory Cohort | Treatment-naive Cohort | Ibrutinib-intolerant Cohort | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort | Ibrutinib Relapsed/Refractory Cohort
Started | 134 | 99 | 33 | 29 | 6
Completed | 41 | 70 | 6 | 3 | 0
Not Completed | 93 | 29 | 27 | 26 | 6
Not completed — Completed 30-Day safety follow-up visit | 53 | 16 | 12 | 2 | 1
Not completed — Death | 13 | 2 | 2 | 11 | 2
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 0
Not completed — Started other anti-cancer therapy | 17 | 4 | 7 | 9 | 3
Not completed — Withdrawal by Subject | 3 | 1 | 1 | 1 | 0
Not completed — Other | 6 | 6 | 4 | 2 | 0

BASELINE CHARACTERISTICS:
Population: All-treated population included all enrolled participants who received 1 or more doses of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Relapsed/Refractory Cohort | Treatment-naive Cohort | Ibrutinib-intolerant Cohort | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort | Ibrutinib Relapsed/Refractory Cohort | Total
Number analyzed (Participants) | 134 | 99 | 33 | 29 | 6 | 301
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.6 (9.2) | 63.5 (9.7) | 63.9 (8.9) | 65.0 (9.6) | 62.5 (7.9) | 64.6 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 33 | 13 | 14 | 3 | 98
  Male | 99 | 66 | 20 | 15 | 3 | 203
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 0 | 0 | 0 | 5
  Not Hispanic or Latino | 129 | 94 | 33 | 28 | 6 | 290
  Unknown or Not Reported | 3 | 2 | 0 | 1 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 1
  Asian | 1 | 2 | 0 | 0 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 2 | 1 | 1 | 15
  White | 120 | 88 | 31 | 27 | 5 | 271
  More than one race | 6 | 4 | 0 | 1 | 0 | 11
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs) in Phase 1
Description: Participants with DLTs in Phase 1 are reported. The DLT was defined as any of the following events unless the adverse event is clearly related to disease progression or the participant's current medical history and associated comorbidities: (1) Any Grade 3 or greater nonhematologic toxicity with the exceptions of alopecia and Grade 3 nausea, vomiting, and diarrhea that respond to supportive therapy; (2) Hematologic toxicities including Grade 4 neutropenia lasting more than 5 days, Grade 4 or Grade 3 thrombocytopenia with bleeding or any requirement for platelets transfusion, Grade 3 or greater febrile neutropenia (body temperature of 38.5 degrees Celsius or more), or Grade 4 anemia, unexplained by underlying disease; or (3) Dosing delay due to toxicity for > 7 consecutive days.
Time Frame: From Day 1 to Day 28 after first dose of study drug
Population: All-treated population included all participants enrolled in Phase 1 (dose-escalation) of the study, received 1 or more doses of study drug, and observed from Day 1 to Day 28 after first dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Participants with CLL/SLL received oral acalabrutinib Dose 1 QD for 28 days.
- Cohort 2a: Participants with CLL/SLL received oral acalabrutinib Dose 2 QD for 28 days.
- Cohort 2b: Participants with CLL/SLL received oral acalabrutinib Dose 2 BID for 28 days.
- Cohort 3: Participants with CLL/SLL received oral acalabrutinib Dose 3 QD for 28 days.
- Cohort 4a; Cohort 4b: Participants with CLL/SLL received oral acalabrutinib Dose 4 QD for 28 days.
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 3 | Cohort 4a | Cohort 4b
Number analyzed (Participants) | 9 | 8 | 29 | 7 | 6 | 6
Participants | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. A serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. The TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: Day 1 through the final data cutoff date (approximately 7 years 6 months)
Population: All-treated population included all enrolled participants who received 1 or more doses of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relapsed/Refractory Cohort | Treatment-naive Cohort | Ibrutinib-intolerant Cohort | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort | Ibrutinib Relapsed/Refractory Cohort
Number analyzed (Participants) | 134 | 99 | 33 | 29 | 6
Participants
  Any TEAEs | 134 | 99 | 33 | 28 | 6
  Any TESAEs | 86 | 50 | 20 | 18 | 3

3. Primary Outcome: Number of Participants With Treatment Emergent Events of Clinical Interest (ECI)
Description: The treatment emergent ECI included the events identified based on preclinical findings, emerging data from clinical studies relating to acalabrutinib, and pharmacological effects of approved Bruton's tyrosine kinase (BTK) inhibitors and reported after the first dose of the study drug.
Time Frame: Day 1 through the final data cutoff date (approximately 7 years 6 months)
Population: All-treated population included all enrolled participants who received 1 or more doses of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relapsed/Refractory Cohort | Treatment-naive Cohort | Ibrutinib-intolerant Cohort | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort | Ibrutinib Relapsed/Refractory Cohort
Number analyzed (Participants) | 134 | 99 | 33 | 29 | 6
Participants
  Atrial fibrillation | 12 | 6 | 4 | 3 | 0
  Ventricular tachyarrhythmias | 2 | 0 | 0 | 0 | 0
  Anemia | 22 | 10 | 4 | 10 | 1
  Neutropenia | 26 | 9 | 5 | 13 | 1
  Other Leukopenia | 2 | 1 | 1 | 0 | 0
  Thrombocytopenia | 10 | 1 | 4 | 4 | 0
  Major hemorrhage | 11 | 8 | 4 | 0 | 1
  Hepatotoxicity | 4 | 4 | 1 | 3 | 0
  Hypertension | 31 | 29 | 7 | 2 | 0
  Infections | 118 | 86 | 25 | 18 | 4
  Interstitial lung disease/Pneumonitis | 1 | 3 | 0 | 0 | 0
  Second primary malignancies, excluding non-melanoma skin | 23 | 14 | 3 | 1 | 0
  Tumor lysis syndrome | 1 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Important Laboratory Abnormalities With Common Terminology Criteria for Adverse Events (CTCAE) Grade 3 or More
Description: Participants with clinically important laboratory abnormalities with CTCAE Grade 3 or more are reported. Laboratory analysis included hematology, clinical chemistry, amylase, lipase, cardiac troponin I, hepatitis B and C testing, and urinalysis. The CTCAE version 4.03 is a descriptive terminology is used for AE reporting. The CTCAE v4.03 displays Grades 1 through 5 with unique clinical descriptions of severity for each AE based on this general guideline: Grade 3 as severe AE, Grade 4 as life-threatening or disabling AE, and Grade 5 as death related to AE.
Time Frame: Day 1 through the final data cutoff date (approximately 7 years 6 months)
Population: All-treated population included all enrolled participants who received 1 or more doses of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relapsed/Refractory Cohort | Treatment-naive Cohort | Ibrutinib-intolerant Cohort | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort | Ibrutinib Relapsed/Refractory Cohort
Number analyzed (Participants) | 134 | 99 | 33 | 29 | 6
Participants
  Hemoglobin, platelets or neutrophils decreased | 72 | 30 | 14 | 19 | 4
  Absolute neutrophil count (decreased) | 57 | 23 | 11 | 13 | 3
  Hemoglobin (decreased) | 17 | 5 | 3 | 8 | 3
  Platelets (decreased) | 20 | 3 | 4 | 5 | 1
  Leukocytes (decreased) | 12 | 2 | 3 | 6 | 0
  Leukocytes (increased) | 29 | 21 | 7 | 0 | 2
  Absolute lymphocyte count (decreased) | 20 | 7 | 2 | 6 | 0
  Absolute lymphocyte count (increased) | 29 | 8 | 7 | 3 | 1
  Urate (increased) | 24 | 15 | 8 | 5 | 2
  Sodium (decreased) | 12 | 5 | 2 | 3 | 0
  Phosphate (decreased) | 9 | 1 | 1 | 1 | 0
  Potassium (increased) | 3 | 5 | 1 | 0 | 0
  Glucose (increased) | 3 | 1 | 3 | 0 | 0
  Alanine aminotransferase (increased) | 3 | 1 | 1 | 1 | 0
  Calcium (increased) | 5 | 0 | 0 | 1 | 0
  Aspartate aminotransferase (increased) | 2 | 2 | 0 | 0 | 0
  Magnesium (increased) | 2 | 2 | 0 | 0 | 0
  Potassium (decreased) | 2 | 1 | 0 | 1 | 0
  Albumin (decreased) | 2 | 1 | 0 | 0 | 0
  Calcium (decreased) | 2 | 0 | 0 | 1 | 0
  Alkaline phosphatase (increased) | 1 | 0 | 0 | 1 | 0
  Amylase (increased) | 2 | 0 | 0 | 0 | 0
  Bilirubin (increased) | 2 | 0 | 0 | 0 | 0
  Creatinine (increased) | 2 | 0 | 0 | 0 | 0
  Lipase (increased) | 1 | 1 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Abnormal Vital Signs Reported as TEAEs
Description: Participants with clinically abnormal vital signs (blood pressure, respiratory rate, pulse rate, or body temperature) reported as TEAEs are reported.
Time Frame: Day 1 through the final data cutoff date (approximately 7 years 6 months)
Population: All-treated population included all enrolled participants who received 1 or more doses of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Relapsed/Refractory Cohort | Treatment-naive Cohort | Ibrutinib-intolerant Cohort | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort | Ibrutinib Relapsed/Refractory Cohort
Number analyzed (Participants) | 134 | 99 | 33 | 29 | 6
Participants
  Tachycardia | 3 | 8 | 2 | 3 | 0
  Bradycardia | 6 | 1 | 0 | 0 | 0
  Pyrexia | 39 | 14 | 10 | 6 | 0
  Hyperpyrexia | 0 | 0 | 0 | 1 | 0
  Hypothermia | 0 | 1 | 0 | 0 | 0
  Procedural hypotension | 0 | 1 | 0 | 0 | 0
  Blood pressure increased | 0 | 1 | 0 | 0 | 0
  Dyspnoea | 27 | 18 | 6 | 3 | 2
  Dyspnoea exertional | 5 | 5 | 1 | 0 | 1
  Hypertension | 30 | 28 | 6 | 1 | 0
  Hypotension | 7 | 12 | 5 | 1 | 2
  Orthostatic hypotension | 0 | 5 | 1 | 0 | 0
  Essential hypertension | 0 | 0 | 1 | 0 | 0
  Hypertensive crisis | 1 | 0 | 0 | 0 | 0
  Malignant hypertension | 0 | 0 | 0 | 1 | 0
  Palpitations | 13 | 4 | 0 | 0 | 0

6. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 6 Hours (AUC0-6) of Acalabrutinib
Description: The AUC0-6 of acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, and 6 hours postdose on Day 1 and Day 8
Population: Pharmacokinetic (PK) population included all participants who complied with the protocol sufficiently and displayed an evaluable PK profile (e.g. exposure to treatment, availability and integrity of measurements, and absence of major protocol violations). 'Number of participants analyzed' denotes the number of participants evaluated for this outcome measure. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Cohort 1: Participants with CLL/SLL received oral acalabrutinib Dose 1 QD for 28 days and later switched to acalabrutinib Dose 1 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 2a: Participants with CLL/SLL received oral acalabrutinib Dose 2 QD for 28 days and later switched to acalabrutinib Dose 1 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 2b: Participants with CLL received oral acalabrutinib Dose 1 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 2c: Participants with CLL received oral acalabrutinib Dose 5 QD (later switched to Dose 1 BID per protocol amendment 6) until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 3: Participants with CLL received oral acalabrutinib Dose 3 QD (later switched to Dose 1 BID per protocol amendment 6) until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 4a: Participants with CLL received oral acalabrutinib Dose 4 QD for 28 days and later switched to acalabrutinib Dose 1 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 4b: Participants with CLL received oral acalabrutinib Dose 5 BID (later switched to Dose 1 BID per protocol amendment 6) until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 7: Treatment-naïve participants with CLL or SLL received oral acalabrutinib Dose 5 QD (later switched to Dose 1 BID per protocol amendment 6) until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 8a: Participants with CLL or SLL and were not tolerating ibrutinib treatment, received oral acalabrutinib Dose 5 QD (which switched to Dose 1 BID per protocol amendment 4) until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 8b: Participants with CLL or SLL and were not tolerating ibrutinib treatment, received oral acalabrutinib Dose 1 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 9: Participants with DLBCLRS or PLL transformation, received oral acalabrutinib Dose 5 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 10: Participants with CLL/SLL and had relapsed/refractory ibrutinib treatment, received oral acalabrutinib Dose 5 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
- Cohort 11: Treatment-naïve participants with CLL/SLL, received oral acalabrutinib Dose 1 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 7 | 24 | 12 | 6 | 6 | 6 | 33 | 3 | 7 | 6 | 5 | 16
hr*ng/mL
  Day 1: number analyzed (Participants) | 8 | 7 | 24 | 12 | 6 | 6 | 6 | 33 | 3 | 6 | 5 | 5 | 16
  Day 1 | 971 (564) | 1250 (836) | 819 (493) | 2170 (1180) | 1880 (1810) | 2960 (1570) | 1950 (487) | 1740 (1540) | 362 (221) | 670 (471) | 1690 (849) | 1100 (590) | 789 (398)
  Day 8: number analyzed (Participants) | 5 | 7 | 22 | 12 | 4 | 5 | 5 | 29 | 1 | 7 | 6 | 5 | 14
  Day 8 | 631 (193) | 1180 (859) | 858 (419) | 1660 (554) | 1750 (518) | 1630 (1050) | 1690 (1090) | 1480 (986) | 2080 (NA) — Standard deviation (SD) was not calculated as only one participant was evaluated at the time of the analysis. | 834 (713) | 1860 (786) | 1250 (1050) | 642 (310)

7. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Last Measurable Concentration (AUC0-last) of Acalabrutinib
Description: The AUC0-last of acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, and 24 hours postdose on Day 1 and Day 8
Population: The PK population included all participants who complied with the protocol sufficiently and displayed an evaluable PK profile (e.g. exposure to treatment, availability and integrity of measurements, and absence of major protocol violations). 'Number of participants analyzed' denotes the number of participants evaluated for this outcome measure. 'Number analyzed' denotes the number of participants evaluated for the specified time point.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Groups:
- Cohort 9: Participants with CLL/SLL received oral acalabrutinib Dose 5 BID until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 8 | 28 | 13 | 7 | 6 | 6 | 37 | 3 | 8 | 10 | 5 | 17
hr*ng/mL
  Day 1 | 1030 (529) | 1270 (775) | 795 (502) | 2280 (1060) | 2030 (1670) | 3430 (1640) | 1950 (487) | 1790 (1470) | 539 (106) | 570 (451) | 1860 (1570) | 1100 (590) | 850 (462)
  Day 8: number analyzed (Participants) | 7 | 7 | 28 | 13 | 7 | 6 | 6 | 37 | 2 | 8 | 9 | 5 | 16
  Day 8 | 729 (380) | 1180 (861) | 850 (660) | 1850 (882) | 2020 (1170) | 1750 (979) | 1560 (1020) | 1400 (929) | 1180 (NA) — The SD could not be derived due to insufficient number of participants were evaluated at the time of the analysis. | 748 (701) | 1710 (669) | 1260 (1060) | 660 (294)

8. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity (AUC0-inf) of Acalabrutinib
Description: The AUC0-inf of Acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, and 24 hours postdose on Day 1 and Day 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 7 | 24 | 11 | 7 | 5 | 6 | 32 | 3 | 6 | 8 | 4 | 15
hr*ng/mL
  Day 1: number analyzed (Participants) | 8 | 7 | 22 | 11 | 7 | 5 | 6 | 32 | 3 | 5 | 6 | 4 | 15
  Day 1 | 1040 (534) | 1320 (827) | 855 (517) | 2440 (1010) | 2050 (1680) | 3250 (1630) | 1970 (495) | 1910 (1530) | 574 (76.3) | 801 (410) | 1770 (776) | 1350 (373) | 940 (430)
  Day 8: number analyzed (Participants) | 6 | 7 | 24 | 9 | 5 | 5 | 4 | 30 | 1 | 6 | 8 | 4 | 15
  Day 8 | 621 (187) | 1200 (865) | 956 (665) | 1990 (1020) | 2360 (1210) | 1750 (1140) | 1780 (1230) | 1540 (973) | 2120 (NA) — The SD could not be calculated as only one participant was evaluated at the time of the analysis. | 963 (728) | 1750 (701) | 1580 (1030) | 652 (298)

9. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Acalabrutinib
Description: The Cmax of Acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, and 24 hours postdose on Day 1 and Day 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 8 | 28 | 13 | 7 | 5 | 6 | 37 | 3 | 8 | 10 | 5 | 16
ng/mL
  Day 1: number analyzed (Participants) | 8 | 8 | 28 | 12 | 7 | 5 | 6 | 37 | 3 | 8 | 10 | 5 | 16
  Day 1 | 685 (475) | 754 (540) | 706 (499) | 1950 (1460) | 1350 (1170) | 1550 (1230) | 1600 (291) | 1390 (1260) | 206 (240) | 554 (500) | 1190 (925) | 727 (436) | 930 (595)
  Day 8: number analyzed (Participants) | 7 | 6 | 27 | 13 | 7 | 5 | 6 | 36 | 2 | 8 | 9 | 4 | 16
  Day 8 | 521 (308) | 805 (757) | 812 (829) | 1350 (809) | 1350 (933) | 902 (638) | 1320 (1540) | 1020 (747) | 939 (NA) — The SD was not calculated due to insufficient number of participants were evaluated at the time of the analysis. | 616 (660) | 1460 (913) | 610 (751) | 633 (449)

10. Primary Outcome: Time of Maximum Plasma Concentration (Tmax) of Acalabrutinib
Description: The Tmax of Acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, and 24 hours postdose on Day 1 and Day 8
Population: as for outcome 7
Measure: Median (Full Range); unit: Hours
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 8 | 28 | 13 | 7 | 5 | 6 | 37 | 3 | 8 | 10 | 5 | 16
Hours
  Day 1: number analyzed (Participants) | 8 | 8 | 28 | 12 | 7 | 5 | 6 | 37 | 3 | 8 | 10 | 5 | 16
  Day 1 | 1.01 [0.417 to 2.00] | 0.917 [0.500 to 3.83] | 0.750 [0.500 to 2.30] | 1.00 [0.250 to 5.92] | 1.00 [0.500 to 1.83] | 1.00 [0.750 to 4.00] | 0.758 [0.250 to 1.08] | 0.783 [0.250 to 2.10] | 1.30 [0.750 to 2.20] | 0.783 [0.500 to 5.83] | 0.992 [0.500 to 4.05] | 1.00 [0.500 to 1.08] | 0.642 [0.483 to 2.00]
  Day 8: number analyzed (Participants) | 7 | 6 | 27 | 13 | 7 | 5 | 6 | 36 | 2 | 8 | 9 | 4 | 16
  Day 8 | 1.05 [0.500 to 1.17] | 0.517 [0.467 to 1.00] | 0.750 [0.450 to 5.75] | 1.03 [0.500 to 2.10] | 1.00 [0.500 to 1.97] | 0.700 [0.500 to 1.95] | 0.758 [0.500 to 2.07] | 0.750 [0.250 to 2.22] | 1.49 [1.08 to 1.90] | 0.908 [0.467 to 2.03] | 1.00 [0.500 to 2.08] | 1.58 [0.467 to 4.08] | 0.533 [0.250 to 1.85]

11. Primary Outcome: Terminal Elimination Half-life (t1/2) of Acalabrutinib
Description: The t1/2 of acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, and 24 hours postdose on Day 1 and Day 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 7 | 24 | 11 | 7 | 5 | 6 | 32 | 3 | 6 | 8 | 4 | 15
Hours
  Day 1: number analyzed (Participants) | 8 | 7 | 22 | 11 | 7 | 5 | 6 | 32 | 3 | 5 | 6 | 4 | 15
  Day 1 | 1.48 (1.50) | 1.44 (1.60) | 0.914 (0.452) | 0.993 (0.303) | 2.89 (3.12) | 3.52 (4.93) | 0.869 (0.0811) | 1.41 (1.73) | 4.83 (3.69) | 0.900 (0.140) | 0.798 (0.0973) | 1.01 (0.209) | 0.781 (0.137)
  Day 8: number analyzed (Participants) | 6 | 7 | 24 | 9 | 5 | 5 | 4 | 30 | 1 | 6 | 8 | 4 | 15
  Day 8 | 1.09 (0.216) | 0.942 (0.107) | 0.995 (0.621) | 0.902 (0.187) | 0.886 (0.131) | 1.38 (0.546) | 1.13 (0.408) | 1.02 (0.454) | 0.914 (NA) — The SD was not calculated as only one participant was evaluated at the time of the analysis. | 1.25 (0.494) | 0.867 (0.289) | 1.67 (1.41) | 0.811 (0.174)

12. Primary Outcome: Terminal Elimination Rate Constant (λz) of Acalabrutinib
Description: The λz of acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, and 24 hours postdose on Day 1 and Day 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: 1/hr
Groups:
- Cohort 2b: Participants with CLL received oral acalabrutinib Dose 1 twice daily until disease progression or per the investigator considered the study treatment to be intolerable or no longer in the participant's best interest.
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 7 | 24 | 11 | 7 | 5 | 6 | 32 | 3 | 6 | 8 | 4 | 15
1/hr
  Day 1: number analyzed (Participants) | 8 | 7 | 22 | 11 | 7 | 5 | 6 | 32 | 3 | 5 | 6 | 4 | 15
  Day 1 | 0.679 (0.276) | 0.750 (0.307) | 0.848 (0.214) | 0.755 (0.209) | 0.502 (0.300) | 0.557 (0.386) | 0.804 (0.0793) | 0.756 (0.292) | 0.373 (0.468) | 0.784 (0.112) | 0.880 (0.114) | 0.706 (0.144) | 0.916 (0.177)
  Day 8: number analyzed (Participants) | 6 | 7 | 24 | 9 | 5 | 5 | 4 | 30 | 1 | 6 | 8 | 4 | 15
  Day 8 | 0.655 (0.132) | 0.744 (0.0866) | 0.793 (0.191) | 0.798 (0.161) | 0.797 (0.128) | 0.578 (0.243) | 0.679 (0.251) | 0.745 (0.174) | 0.758 (NA) — The SD was not calculated as only one participant was evaluated at the time of the analysis. | 0.623 (0.218) | 0.857 (0.209) | 0.603 (0.324) | 0.894 (0.204)

13. Primary Outcome: Apparent Oral Clearance (CL/F) of Acalabrutinib
Description: The CL/F of acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, and 24 hours postdose on Day 1 and Day 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 7 | 24 | 11 | 7 | 5 | 6 | 32 | 3 | 6 | 8 | 4 | 15
L/hr
  Day 1: number analyzed (Participants) | 8 | 7 | 22 | 11 | 7 | 5 | 6 | 32 | 3 | 5 | 6 | 4 | 15
  Day 1 | 114 (44.4) | 193 (121) | 212 (302) | 112 (98.4) | 265 (263) | 169 (123) | 108 (32.0) | 315 (488) | 352 (43.7) | 311 (166) | 142 (88.9) | 156 (40.3) | 137 (77.4)
  Day 8: number analyzed (Participants) | 6 | 7 | 24 | 9 | 5 | 5 | 4 | 30 | 1 | 6 | 8 | 4 | 15
  Day 8 | 176 (62.1) | 216 (154) | 162 (141) | 122 (55.5) | 131 (70.3) | 344 (242) | 191 (180) | 389 (1070) | 94.5 (NA) — The SD was not calculated as only one participant was evaluated at the time of the analysis. | 336 (258) | 132 (51.8) | 167 (95.1) | 188 (92.5)

14. Primary Outcome: Apparent Volume of Distribution (Vz/F) of Acalabrutinib
Description: The Vz/F of acalabrutinib is reported.
Time Frame: Predose and at 0.25, 0.5, 0.75, 1, 2, 4, 6, and 24 hours postdose on Day 1 and Day 8
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 8a | Cohort 8b | Cohort 9 | Cohort 10 | Cohort 11
Number analyzed (Participants) | 8 | 7 | 24 | 11 | 7 | 5 | 6 | 32 | 3 | 6 | 8 | 4 | 15
L
  Day 1: number analyzed (Participants) | 8 | 7 | 22 | 11 | 7 | 5 | 6 | 32 | 3 | 5 | 6 | 4 | 15
  Day 1 | 268 (332) | 574 (992) | 450 (1250) | 182 (230) | 2100 (3290) | 1480 (2850) | 133 (30.0) | 930 (1750) | 2600 (2030) | 422 (290) | 171 (125) | 235 (105) | 158 (102)
  Day 8: number analyzed (Participants) | 6 | 7 | 24 | 9 | 5 | 5 | 4 | 30 | 1 | 6 | 8 | 4 | 15
  Day 8 | 286 (150) | 302 (238) | 333 (729) | 165 (104) | 172 (114) | 739 (745) | 384 (466) | 1180 (4940) | 125 (NA) — The SD was not calculated as only one participant was evaluated at the time of the analysis. | 726 (814) | 179 (134) | 533 (716) | 234 (162)

15. Secondary Outcome: Percentage of Participants With Objective Response (OR) as Assessed by the Investigator
Description: For CLL/SLL, OR is defined as complete remission (CR), CR with incomplete marrow recovery (CRi), or partial remission (PR). CR: lymphocytes (lympho) <4×10^9/L, normocellular bone marrow (BM), normal lymph nodes (NLN), liver and spleen (L/S), absolute neutrophil count (ANC) >1.5×10^9/L, platelets >100×10^9/L, hemoglobin (Hb) >11g/dL. Cri: lympho <4×10^9/L, hypocellular BM, NLN, L/S, persistent anemia, hrombocytopenia, or neutropenia. PR: >=50% reduction in lymphadenopathy and/or enlargement of L/S or lympho (<5×10^9/L or >=50% decrease from baseline) and criteria of ANC/platelets/Hb per CR or >=50% improvement over baseline. Hematology result were without exogenous growth factors/transfusion. For RS, OR as CR or PR by Cheson et al. 2014 based on PET/CT scans and bone marrow. CR: disappearance of all detectable clinical evidence of disease and disease-related symptoms and PR: >=50% decrease in sum of the product diameter of 6 largest nodal masses and no new sites of disease.
Time Frame: Day 1 through the final data cutoff date (approximately 7 years 6 months)
Population: Efficacy evaluable population included all enrolled participants who received 1 or more doses of study drug and had 1 or more response assessments after the first dose of study drug.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 11
Number analyzed (Participants) | 8 | 8 | 63 | 32 | 7 | 6 | 6 | 37 | 60
Percentage of participants | 100.0 [63.1 to 100.0] | 75 [34.9 to 96.8] | 92.1 [82.4 to 97.4] | 93.8 [79.2 to 99.2] | 100.0 [59.0 to 100.0] | 100.0 [54.1 to 100.0] | 100.0 [54.1 to 100.0] | 97.3 [85.8 to 99.9] | 100.0 [94.0 to 100.0]

16. Secondary Outcome: Duration of Response (DOR) as Assessed by the Investigator
Description: The DoR is defined as the time from the date of achieving the first CR, CRi, or PR to the date of progressive disease (PD) or death due to any cause, whichever occurred first. The CR, CRi, or PR are defined in the above outcome measure. For CLL/SLL, PD is defined as lympho >=50% increase from baseline with >= 5000 B lymphocytes/µL, progressive cytopenias by bone marrow biopsy, appearance of any new lesion or new appearance of hepatomegaly or splenomegaly or >= 50 % increase in lymphadenopathy/hepatomegaly/splenomegaly, platelets decrease of >=50% from baseline secondary to CLL or < 100,000/µL and worsening bone marrow or Hb decrease of > 2 g/dL from baseline secondary to CLL or decrease to less than 100 g/L and worsening bone marrow. For RS, PD is defined as an increase by 25 % in longest diameter, new lesion or assessable disease progression. The DoR was estimated using Kaplan-Meier method.
Time Frame: Day 1 through the final data cutoff date (approximately 7 years 6 months)
Population: Efficacy evaluable population included all enrolled participants who received 1 or more doses of study drug and had 1 or more response assessments after the first dose of study drug. The DoR was analyzed for participants who achieved OR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 11
Number analyzed (Participants) | 8 | 6 | 58 | 30 | 7 | 6 | 6 | 36 | 60
Months | 33.3 [13.8 to NA] — Upper limit of 95% confidence interval (CI) was not calculated because insufficient number of participants had DoR. | 26.7 [13.9 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had DoR. | 77.3 [46.3 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had DoR. | 43.0 [29.4 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had DoR. | NA [9.0 to NA] — Median and upper limit of 95% CI were not calculated because insufficient number of participants had DoR. | 64.1 [19.4 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had DoR. | NA [38.9 to NA] — Median and upper limit of 95% CI were not calculated because insufficient number of participants had DoR. | NA [NA to NA] — Median and 95% CI were not calculated because insufficient number of participants had DoR. | NA [NA to NA] — Median and 95% CI were not calculated because insufficient number of participants had DoR.

17. Secondary Outcome: Progression Free Survival (PFS) as Assessed by the Investigator
Description: The PFS is defined as the time from the date of first dose of study drug to the date of first PD or death due to any cause, whichever occurred first. For CLL/SLL, PD is defined as lympho >= 50 % increase from baseline with >= 5000 B lymphocytes/µL, progressive cytopenias by bone marrow biopsy, appearance of any new lesion or new appearance of hepatomegaly or splenomegaly or >= 50 % increase in lymphadenopathy/hepatomegaly/splenomegaly, platelets decrease of >= 50 % from baseline secondary to CLL or < 100,000/µL and worsening bone marrow or Hb decrease of > 2 g/dL from baseline secondary to CLL or decrease to less than 100 g/L and worsening bone marrow. For RS, PD is defined as an increase by 25 % in longest diameter, new lesion or assessable disease progression. The PFS was estimated using Kaplan-Meier method.
Time Frame: Day 1 through the final data cutoff date (approximately 7 years 6 months)
Population: as for outcome 15
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 | Cohort 2a | Cohort 2b | Cohort 2c | Cohort 3 | Cohort 4a | Cohort 4b | Cohort 7 | Cohort 11
Number analyzed (Participants) | 9 | 8 | 65 | 33 | 7 | 6 | 6 | 37 | 62
Months | 38.3 [15.5 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had PFS. | 33.1 [15.8 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had PFS. | 79.1 [49.8 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had PFS. | 46.6 [33.9 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had PFS. | NA [12.7 to NA] — Median and upper limit of 95% CI were not calculated because insufficient number of participants had PFS.. | 67.8 [33.2 to NA] — Upper limit of 95% CI was not calculated because insufficient number of participants had PFS. | NA [40.7 to NA] — Median and upper limit of 95% CI were not calculated because insufficient number of participants had PFS.. | NA [NA to NA] — Median and 95% CI were not calculated because insufficient number of participants had PFS.. | NA [NA to NA] — Median and 95% CI were not calculated because insufficient number of participants had PFS..

ADVERSE EVENTS:
Time Frame: Day 1 through the final data cutoff date (approximately 7 years 6 months)
Arm/Group | Relapsed/Refractory Cohort | Treatment-naive Cohort | Ibrutinib-intolerant Cohort | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort | Ibrutinib Relapsed/Refractory Cohort
All-Cause Mortality (participants affected / at risk) | 13/134 | 2/99 | 2/33 | 11/29 | 2/6
Serious Adverse Events (participants affected / at risk) | 86/134 | 50/99 | 20/33 | 18/29 | 3/6
Other Adverse Events (participants affected / at risk) | 134/134 | 99/99 | 33/33 | 28/29 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed/Refractory Cohort (N=134) | Treatment-naive Cohort (N=99) | Ibrutinib-intolerant Cohort (N=33) | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort (N=29) | Ibrutinib Relapsed/Refractory Cohort (N=6)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epiploic appendagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Methaemoglobinaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Splenic infarction (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Infusion site injury (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Perforation bile duct (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Brain abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Bronchitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 pneumonia (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytomegalovirus infection reactivation (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis rotavirus (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella bacteraemia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycobacterium avium complex infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 19 (24) | 6 (8) | 3 (8) | 1 (1) | 0 (0)
Pneumonia fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (2) | 1 (2) | 3 (3) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pseudomonal sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (6) | 2 (3) | 0 (0) | 2 (2) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (6) | 2 (6) | 2 (2) | 0 (0) | 0 (0)
Viral myocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cytomegalovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immunosuppressant drug level increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin i increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angiosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Benign lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Central nervous system leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuroendocrine carcinoma of the skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plasmablastic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Multiple system atrophy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 5 (5) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Relapsed/Refractory Cohort (N=134) | Treatment-naive Cohort (N=99) | Ibrutinib-intolerant Cohort (N=33) | Richters Syndrome/Prolymphocytic Leukemia Transformation Cohort (N=29) | Ibrutinib Relapsed/Refractory Cohort (N=6)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 5 (6) | 5 (6) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 29 (39) | 28 (60) | 6 (8) | 1 (1) | 0 (0)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 7 (7) | 11 (11) | 5 (6) | 1 (1) | 2 (2)
Lymphoedema (Vascular disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 5 (7) | 1 (1) | 0 (0) | 0 (0)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Eyelid thickening (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Plethoric face (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poor peripheral circulation (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 3 (3) | 1 (2) | 0 (0) | 0 (0)
Metamorphopsia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night blindness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular hypertension (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Posterior capsule opacification (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal artery occlusion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Retinal haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Retinal tear (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Strabismus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 5 (6) | 9 (9) | 0 (0) | 1 (1) | 0 (0)
Visual acuity reduced (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 7 (7) | 6 (6) | 3 (3) | 1 (1) | 0 (0)
Vitreous degeneration (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 11 (12) | 8 (8) | 3 (3) | 2 (2) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 16 (24) | 10 (17) | 3 (4) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 11 (12) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal fissure haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 3 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Barrett's oesophagus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath odour (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coeliac disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 35 (41) | 20 (22) | 7 (9) | 2 (2) | 1 (1)
Dental caries (Gastrointestinal disorders) | 11 (13) | 5 (6) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 71 (131) | 53 (93) | 20 (31) | 14 (19) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Dumping syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 14 (14) | 10 (11) | 6 (6) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 9 (9) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eosinophilic oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 7 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (12) | 17 (20) | 2 (2) | 1 (1) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gingival blister (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival discolouration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia teeth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 21 (42) | 8 (14) | 4 (8) | 7 (9) | 1 (1)
Large intestinal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip dry (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lip erythema (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 2 (3) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 47 (67) | 34 (53) | 11 (16) | 4 (4) | 2 (2)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 18 (27) | 9 (12) | 4 (7) | 9 (13) | 1 (2)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral blood blister (Gastrointestinal disorders) | 5 (5) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Oral disorder (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oral mucosa haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 5 (5) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Peritoneal haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 2 (4) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (17) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Pseudopolyposis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal discharge (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 3 (4) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Rectal polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spigelian hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 13 (16) | 14 (23) | 5 (6) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue geographic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tongue haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 6 (8) | 7 (8) | 1 (1) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 33 (44) | 24 (30) | 9 (12) | 3 (3) | 1 (1)
Asthenia (General disorders) | 6 (7) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Axillary pain (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Catheter site haemorrhage (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 4 (5) | 3 (4) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 16 (18) | 13 (14) | 3 (3) | 2 (3) | 1 (1)
Complication associated with device (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Crepitations (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Face oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial pain (General disorders) | 1 (1) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Fat necrosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 49 (58) | 22 (31) | 7 (10) | 6 (8) | 1 (1)
Feeling cold (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Granuloma (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hernia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 12 (14) | 13 (14) | 2 (3) | 1 (1) | 0 (0)
Infusion site rash (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site bruising (General disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Injection site phlebitis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malaise (General disorders) | 6 (7) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Medical device site bruise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 8 (11) | 12 (16) | 8 (8) | 3 (3) | 0 (0)
Oedema (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 28 (36) | 18 (25) | 7 (7) | 2 (2) | 0 (0)
Pain (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 4 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Physical deconditioning (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyp (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 39 (69) | 13 (19) | 10 (17) | 6 (12) | 0 (0)
Suprapubic pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Swelling face (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Systemic inflammatory response syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site mass (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 10 (11) | 5 (8) | 2 (2) | 3 (6) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic mass (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod bite (Immune system disorders) | 7 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Allergy to arthropod sting (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contrast media allergy (Immune system disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Graft versus host disease in skin (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypogammaglobulinaemia (Immune system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Immunodeficiency (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspergillus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body tinea (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 14 (18) | 14 (16) | 6 (9) | 2 (3) | 0 (0)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Burkholderia cepacia complex infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 4 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Campylobacter infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 12 (13) | 1 (1) | 3 (7) | 0 (0) | 0 (0)
Chronic sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 3 (3) | 0 (0)
Bradycardia (Cardiac disorders) | 5 (8) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccidioidomycosis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 7 (7) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 7 (8) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Bundle branch block left (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epstein-barr virus infection reactivation (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye infection (Infections and infestations) | 4 (5) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fungal infection (Infections and infestations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fungal skin infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Furuncle (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 6 (7) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Infected bite (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infected dermal cyst (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 12 (13) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 9 (12) | 1 (1) | 3 (5) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphangitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metapneumovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Moraxella infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mycobacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myringitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nail infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 11 (12) | 9 (11) | 3 (6) | 0 (0) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Oral herpes (Infections and infestations) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 6 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 26 (29) | 12 (16) | 3 (9) | 3 (3) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-acute covid-19 syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Propionibacterium infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Prostatic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomonas infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 4 (4) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Salmonellosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 33 (44) | 22 (34) | 3 (6) | 2 (3) | 1 (1)
Sinusitis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea cruris (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinea versicolour (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 3 (4) | 6 (6) | 2 (3) | 0 (0) | 0 (0)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 54 (88) | 49 (85) | 15 (25) | 3 (3) | 1 (1)
Ureteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 15 (32) | 13 (24) | 5 (11) | 2 (2) | 0 (0)
Mitral valve disease (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection enterococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular device infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anaemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 10 (10) | 8 (13) | 1 (1) | 0 (0) | 0 (0)
Axillary web syndrome (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chest injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 42 (60) | 50 (62) | 11 (13) | 5 (6) | 0 (0)
Palpitations (Cardiac disorders) | 13 (15) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dental restoration failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 21 (41) | 23 (34) | 6 (11) | 4 (4) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fractured coccyx (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 5 (6) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Human bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 5 (6) | 10 (11) | 1 (1) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 4 (4) | 4 (5) | 1 (1) | 1 (1) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Muscle rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 5 (5) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural inflammation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural swelling (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural hypotension (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Reactive gastropathy (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Scrotal haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 2 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 6 (7) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Skin wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 3 (3) | 8 (9) | 2 (2) | 3 (3) | 0 (0)
Stoma site reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomal hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 6 (9) | 8 (12) | 0 (0) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Venous injury (Injury, poisoning and procedural complications) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (4) | 0 (0) | 2 (2) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Antinuclear antibody positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (4) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Bk polyomavirus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood albumin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood beta-d-glucan increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 7 (9) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Blood folate decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood immunoglobulin g decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood sodium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood testosterone decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone density decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 1 (1) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Coagulation time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Computerised tomogram thorax abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eastern cooperative oncology group performance status worsened (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram qt prolonged (Investigations) | 1 (1) | 1 (3) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza a virus test positive (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza b virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Influenza virus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (3) | 0 (0) | 0 (0) | 3 (6) | 0 (0)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Norovirus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 4 (7) | 0 (0) | 1 (8) | 4 (4) | 0 (0)
Prostatic specific antigen increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngocele (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid hormones increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin i increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin increased (Investigations) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 27 (43) | 8 (13) | 3 (5) | 4 (6) | 0 (0)
Weight increased (Investigations) | 34 (97) | 33 (105) | 10 (22) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 22 (26) | 13 (19) | 2 (2) | 4 (4) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 4 (5) | 7 (7) | 2 (3) | 3 (3) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Porokeratosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypernatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphagia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 4 (4) | 6 (6) | 1 (2) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 2 (3) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (8) | 4 (4) | 0 (0) | 4 (5) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b complex deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin b12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin d deficiency (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 (78) | 55 (83) | 9 (13) | 6 (8) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 7 (8) | 10 (10) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 19 (21) | 22 (26) | 3 (3) | 4 (5) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 3 (4) | 2 (2) | 0 (0)
Bursa disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 3 (3) | 2 (2) | 1 (2) | 0 (0) | 0 (0)
Joint hyperextension (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb mass (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medial tibial stress syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 11 (14) | 14 (20) | 3 (4) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 (6) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (22) | 14 (17) | 8 (10) | 3 (3) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteopenia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 5 (5) | 6 (6) | 2 (2) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 24 (32) | 11 (14) | 5 (7) | 4 (4) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus tarsi syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Trigger finger (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vertebral column mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (12) | 11 (17) | 4 (4) | 0 (0) | 0 (0)
Basosquamous carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of urethra (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukaemia cutis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 15 (15) | 10 (10) | 3 (3) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 3 (3) | 6 (6) | 1 (1) | 1 (1) | 0 (0)
Sebaceous adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 (6) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Sinonasal papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Skin neoplasm bleeding (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (9) | 7 (7) | 1 (1) | 0 (0) | 0 (0)
Tongue neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Middle ear effusion (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Carotid arteriosclerosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery aneurysm (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Motion sickness (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral microhaemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cognitive disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dementia alzheimer's type (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 24 (27) | 20 (22) | 6 (7) | 4 (6) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 4 (4) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 68 (98) | 48 (79) | 14 (18) | 12 (16) | 1 (3)
Hemianopia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypersomnia (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Hypogeusia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Idiopathic partial epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intracranial pressure increased (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 5 (6) | 5 (6) | 2 (3) | 0 (0) | 0 (0)
Mental impairment (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 8 (9) | 4 (4) | 5 (6) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 19 (19) | 14 (15) | 5 (5) | 1 (2) | 0 (0)
Parosmia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (5) | 5 (5) | 2 (2) | 2 (2) | 0 (0)
Post herpetic neuralgia (Nervous system disorders) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 6 (7) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Resting tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Retinal migraine (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 6 (7) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Sinus headache (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Spinal cord disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 6 (6) | 7 (9) | 2 (2) | 0 (0) | 0 (0)
Taste disorder (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Anger (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 14 (15) | 9 (12) | 2 (2) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (4) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Depressed mood (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 10 (10) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Emotional distress (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 18 (20) | 19 (20) | 5 (5) | 4 (4) | 0 (0)
Libido decreased (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Phonophobia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Premature ejaculation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 7 (9) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Bladder hypertrophy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 3 (6) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 6 (8) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 7 (8) | 10 (13) | 3 (3) | 1 (1) | 0 (0)
Lower urinary tract symptoms (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 6 (6) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 7 (9) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Thyroid calcification (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 9 (9) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 18 (20) | 8 (8) | 3 (4) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal mass (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcapsular renal haematoma (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urge incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid disorder (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 5 (5) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 4 (4) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 4 (4) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 5 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Genital haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Thyroid mass (Endocrine disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Penile oedema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peyronie's disease (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostatic obstruction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 7 (9) | 6 (7) | 1 (1) | 0 (0) | 0 (0)
Scrotal haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Testicular mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acquired diaphragmatic eventration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract nuclear (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Asthma exercise induced (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 47 (63) | 32 (41) | 13 (19) | 4 (12) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 27 (36) | 17 (18) | 6 (6) | 3 (3) | 2 (2)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 5 (5) | 1 (1) | 0 (0) | 1 (1)
Chorioretinopathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 (25) | 12 (19) | 4 (7) | 3 (3) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (6) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 20 (30) | 28 (30) | 6 (7) | 1 (1) | 0 (0)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 (26) | 17 (22) | 4 (4) | 0 (0) | 0 (0)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (6) | 1 (1) | 5 (6) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 20 (28) | 8 (9) | 3 (5) | 2 (2) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dacryostenosis acquired (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 13 (15) | 14 (14) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 16 (17) | 9 (10) | 1 (2) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 5 (5) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 6 (6) | 0 (0) | 0 (0) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tonsillolith (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Jaundice acholuric (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Episcleritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 11 (16) | 5 (5) | 0 (0) | 0 (0)
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 10 (11) | 5 (5) | 2 (4) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (9) | 8 (8) | 1 (1) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Brachioradial pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermal cyst (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 13 (14) | 6 (7) | 6 (7) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 17 (18) | 16 (17) | 5 (5) | 0 (0) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5) | 3 (3) | 0 (0) | 0 (0)
Eczema nummular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 12 (12) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Erythema annulare (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Follicular mucinosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye inflammation (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Granulomatous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hand dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 12 (14) | 11 (14) | 2 (2) | 2 (2) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macule (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Madarosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nail bed bleeding (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail bed inflammation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail ridging (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Necrobiosis lipoidica diabeticorum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 21 (24) | 15 (19) | 2 (3) | 2 (2) | 0 (0)
Eye movement disorder (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodular rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panniculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 28 (34) | 18 (24) | 3 (3) | 2 (2) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Poikiloderma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (4) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (15) | 8 (10) | 2 (2) | 2 (3) | 0 (0)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Purpura senile (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 21 (23) | 18 (23) | 6 (6) | 2 (2) | 1 (1)
Rash erythematous (Skin and subcutaneous tissue disorders) | 6 (6) | 4 (5) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 17 (18) | 12 (13) | 3 (4) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rosacea (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin fragility (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 18 (22) | 5 (5) | 5 (5) | 0 (0) | 0 (0)
Skin mass (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (5) | 3 (3) | 0 (0) | 0 (0)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Solar lentigo (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (6) | 3 (3) | 1 (1) | 0 (0) | 1 (1)
Excessive exercise (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm (Vascular disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Eyelid pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachiocephalic vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Capillary disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Essential hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extravasation blood (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 6 (6) | 5 (6) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The Phase 2 dose was chosen on the basis of the pharmacodynamics data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT02029443/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-25): https://cdn.clinicaltrials.gov/large-docs/43/NCT02029443/SAP_001.pdf